CLINICAL TRIAL: NCT00231985
Title: Behavior Therapy and Psychosocial Treatment for Tourette Syndrome and Chronic Tic Disorder
Brief Title: Effectiveness of Behavior Therapy and Psychosocial Therapy for the Treatment of Tourette Syndrome and Chronic Tic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH069877 (NIH); R01MH069877 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Tourette Syndrome; Tic Disorders
Keywords: Habit-reversal Therapy; Behavior Therapy; Supportive Therapy
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator): Participants will receive supportive psychotherapy.
  Interventions: Behavioral: Supportive therapy
- 2 (Active Comparator): Participants will receive habit reversal therapy.
  Interventions: Behavioral: Habit reversal therapy

INTERVENTIONS:
Behavioral: Habit reversal therapy — Habit reversal therapy consists of awareness training, relaxation training, self-monitoring, and competing response training.
  Arms: 2
Behavioral: Supportive therapy — Supportive therapy focuses on educating participants about tics: how tics present themselves, the causes of tics, the common conditions that may occur along with tics, and environmental factors that may affect their tics (e.g. family, social, school, stress).
  Arms: 1

SUMMARY:
This study will compare the efficacy of supportive therapy versus habit-reversal therapy for the treatment of Tourette syndrome and chronic tic disorder.

DETAILED DESCRIPTION:
Tourette syndrome and chronic tic disorder are neurological disorders characterized by tics. Tics are involuntary, rapid motor movements or vocalizations that occur suddenly and repeatedly. In adults, the symptoms of Tourette syndrome or chronic tic disorder can be severe. These symptoms often cause difficulties in interpersonal relationships and high unemployment rates. Medication treatments are available for both Tourette syndrome and chronic tic disorder, but most are not completely effective and cause considerable negative side effects. Therefore, non-medication treatments are needed. This study will compare the efficacy of supportive therapy versus habit-reversal therapy for the treatment of Tourette syndrome and chronic tic disorder.

Participants in this open-label study will be randomly assigned to receive either supportive therapy or habit-reversal therapy. Over the course of 10 weeks, all participants will receive 8 treatment sessions of their assigned therapy. The supportive therapy will focus on educating participants on what tics are, how tics present themselves, the causes of tics, the common conditions that may occur along with tics, and environmental factors that may affect their tics (e.g. family, social, school, stress). Habit-reversal therapy will consist of awareness training, relaxation training, self-monitoring, and competing response training. Tic severity, tic-related impairment, depressive symptoms, anxiety symptoms, and obsessive-compulsive symptoms will be assessed at each study session, using diagnostic interviews and self-report scales.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for Tourette syndrome or chronic tic disorder
* The primary reason for seeking treatment is Tourette syndrome and/or chronic tic disorder
* Either Tourette syndrome or chronic tic disorder is of more concern than any other simultaneous disease or disorder
* Score greater than 3 on the Clinical Global Impressions Severity Scale
* Score greater than 14 on the Yale Global Tic Severity Scale
* Unmedicated or on stable medication treatment for tics, obsessive compulsive disorder, attention deficit hyperactivity disorder, and/or depressive disorder for at least 6 weeks, and not planning to change medication for the duration of study participation

Exclusion Criteria:

* Total tic score greater than 33
* Score less than 80 on the Wechsler Test of Adult Reading
* DSM-IV diagnosis of alcohol or substance dependence within the 3 months prior to study enrollment
* Currently taking psychotropic medications for any psychiatric disorder (except for tics, obsessive compulsive disorder, attention deficit hyperactivity disorder, and/or depressive disorder)
* Any serious psychiatric disorder (e.g., bipolar disorder, psychosis) that requires immediate alternative treatment
* Previously treated with four or more sessions of habit-reversal therapy for tics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Tic severity | Measured at Week 10

SECONDARY OUTCOMES:
Tic-related impairment | Measured at Week 10
Depressive symptoms | Measured at Week 10
Anxiety symptoms | Measured at Week 10
Obsessive-compulsive symptoms | Measured at Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — MGH/Harvard Medical School
Locations (3):
- United States (3):
  - Yale Child Study Center, Yale University, New Haven, Connecticut
  - OCD Clinic/Psychiatry, Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas Health Sciences Center, San Antonio, Texas

REFERENCES:
- [Background] Lin H, Yeh CB, Peterson BS, Scahill L, Grantz H, Findley DB, Katsovich L, Otka J, Lombroso PJ, King RA, Leckman JF. Assessment of symptom exacerbations in a longitudinal study of children with Tourette's syndrome or obsessive-compulsive disorder. J Am Acad Child Adolesc Psychiatry. 2002 Sep;41(9):1070-7. doi: 10.1097/00004583-200209000-00007. PMID 12218428
- [Background] Bruun RD. Subtle and underrecognized side effects of neuroleptic treatment in children with Tourette's disorder. Am J Psychiatry. 1988 May;145(5):621-4. doi: 10.1176/ajp.145.5.621. PMID 2895987
- [Background] Scahill L, Chappell PB, King RA, Leckman JF. Pharmacologic treatment of tic disorders. Child Adolesc Psychiatr Clin N Am. 2000 Jan;9(1):99-117. PMID 10674192
- [Derived] Weingarden H, Scahill L, Hoeppner S, Peterson AL, Woods DW, Walkup JT, Piacentini J, Wilhelm S. Self-esteem in adults with Tourette syndrome and chronic tic disorders: The roles of tic severity, treatment, and comorbidity. Compr Psychiatry. 2018 Jul;84:95-100. doi: 10.1016/j.comppsych.2018.04.008. Epub 2018 Apr 23. PMID 29729555
- [Derived] Houghton DC, Capriotti MR, Scahill LD, Wilhelm S, Peterson AL, Walkup JT, Piacentini J, Woods DW. Investigating Habituation to Premonitory Urges in Behavior Therapy for Tic Disorders. Behav Ther. 2017 Nov;48(6):834-846. doi: 10.1016/j.beth.2017.08.004. Epub 2017 Aug 10. PMID 29029679
- [Derived] Sukhodolsky DG, Woods DW, Piacentini J, Wilhelm S, Peterson AL, Katsovich L, Dziura J, Walkup JT, Scahill L. Moderators and predictors of response to behavior therapy for tics in Tourette syndrome. Neurology. 2017 Mar 14;88(11):1029-1036. doi: 10.1212/WNL.0000000000003710. Epub 2017 Feb 15. PMID 28202705
- [Derived] Peterson AL, McGuire JF, Wilhelm S, Piacentini J, Woods DW, Walkup JT, Hatch JP, Villarreal R, Scahill L. An Empirical Examination of Symptom Substitution Associated With Behavior Therapy for Tourette's Disorder. Behav Ther. 2016 Jan;47(1):29-41. doi: 10.1016/j.beth.2015.09.001. Epub 2015 Sep 11. PMID 26763495
- [Derived] McGuire JF, Piacentini J, Scahill L, Woods DW, Villarreal R, Wilhelm S, Walkup JT, Peterson AL. Bothersome tics in patients with chronic tic disorders: Characteristics and individualized treatment response to behavior therapy. Behav Res Ther. 2015 Jul;70:56-63. doi: 10.1016/j.brat.2015.05.006. Epub 2015 May 12. PMID 25988365
- [Derived] McGuire JF, Nyirabahizi E, Kircanski K, Piacentini J, Peterson AL, Woods DW, Wilhelm S, Walkup JT, Scahill L. A cluster analysis of tic symptoms in children and adults with Tourette syndrome: clinical correlates and treatment outcome. Psychiatry Res. 2013 Dec 30;210(3):1198-204. doi: 10.1016/j.psychres.2013.09.021. Epub 2013 Sep 27. PMID 24144615
- [Derived] Jeon S, Walkup JT, Woods DW, Peterson A, Piacentini J, Wilhelm S, Katsovich L, McGuire JF, Dziura J, Scahill L. Detecting a clinically meaningful change in tic severity in Tourette syndrome: a comparison of three methods. Contemp Clin Trials. 2013 Nov;36(2):414-20. doi: 10.1016/j.cct.2013.08.012. Epub 2013 Aug 31. PMID 24001701
- [Derived] Wilhelm S, Peterson AL, Piacentini J, Woods DW, Deckersbach T, Sukhodolsky DG, Chang S, Liu H, Dziura J, Walkup JT, Scahill L. Randomized trial of behavior therapy for adults with Tourette syndrome. Arch Gen Psychiatry. 2012 Aug;69(8):795-803. doi: 10.1001/archgenpsychiatry.2011.1528. PMID 22868933
- See also: Click here for the Tourette Syndrome Association Web site — http://tsa-usa.org
- See also: Click here for the Tic Disorders Clinic & Research Unit at the Massachusetts General Hospital/Harvard Medical School — http://www.mghocd.org/tics
- See also: Click here for the TS/OCD Specialty Clinic at the Yale Child Study Center — http://info.med.yale.edu/chldstdy/tsocd/